CLINICAL TRIAL: NCT01201356
Title: A Single Arm, Open-label, Multicenter Study Evaluating the Long-term Safety and Tolerability of 0.5 mg Fingolimod (FTY720) Administered Orally Once Daily in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: Long-term Safety and Tolerability of 0.5 mg Fingolimod in Patients With Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720D2399; 2010-020515-37 (EudraCT Number)
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Results first posted 2019-11-07 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Relapsing Forms of Multiple Sclerosis
Keywords: Fingolimod; FTY720; Relapsing forms of MS; Multiple Sclerosis; Efficacy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fingolimod 0.5 mg/day (Experimental): Open-label fingolimod 0.5 mg, taken orally once daily
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — 0.5 mg/day
  Other Names: FTY720

SUMMARY:
The purpose of this study was to collect long-term safety and tolerability, long-term efficacy, and health outcome data in all patients currently ongoing in the fingolimod multiple sclerosis clinical development program. This study combined all currently ongoing Phase II and III fingolimod extension studies as well as ongoing and newly planned studies into one single long-term extension protocol that provided patients with continuous treatment until fingolimod was registered, commercially available, and reimbursed in the respective countries.

DETAILED DESCRIPTION:
This study had two parts:

* Part 1, collecting long-term safety, tolerability, efficacy and health outcomes data through approximately 30-Jun-2016 until all end of study (EOS) visits of Part 1 and last follow-up visit through Jan-2017 and
* Part 2, collecting limited safety and tolerability data until approximately 30 Jun 2018, in a subset of patients who participated in Part 1, and other eligible patients from ongoing fingolimod trials.

ELIGIBILITY:
Key Inclusion Criteria:

- Patients who have completed selected ongoing or planned trials with FTY720.

Key Exclusion Criteria:

* Premature permanent discontinuation of a previous fingolimod study.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, UNLESS they are using two birth control methods, at least 1 of which must be hormonal contraception, tubal sterilization, partner's vasectomy or intrauterine device.
* Chronic disease of the immune system, other than multiple sclerosis, which may require immunosuppressive treatment.
* Diabetic patients with moderate or severe non-proliferative diabetic retinopathy or proliferative diabetic retinopathy and uncontrolled diabetic patients with HbA1c > 8%.
* Active systemic bacterial, viral or fungal infections, or known to have AIDS, Hepatitis B, Hepatitis C infection or have positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody tests.
* Previous treatment with cladribine, cyclophosphamide or mitoxantrone.
* Treatment with immunoglobulins and/or monoclonal antibodies (including Natalizumab) in the past 3 months during the previous fingolimod study:
* Any of the following cardiovascular conditions that have developed during the previous fingolimod study:

  * Myocardial infarction within the past 6 months prior to entry in the extension study or with current unstable ischemic heart disease;
  * Cardiac failure (Class III, according to New York Heart Association Classification) or any severe cardiac disease as determined by the investigator;
  * Arrhythmia requiring current treatment with Class III antiarrhythmic drugs (e.g., amiodarone, bretylium, sotalol, ibutilide, azimilide, dofetilide)
  * History or presence of a third degree AV block
  * Proven history of sick sinus syndrome or sino-atrial heart block
  * Known history of angina pectoris due to coronary spasm or Raynaud's phenomenon
* Any of the following pulmonary conditions during the previous fingolimod study:

  * Severe respiratory disease or pulmonary fibrosis diagnosed (during the previous fingolimod study)
  * Active tuberculosis
* Alcohol abuse, chronic liver disease during the previous fingolimod study.

The patient must have participated in a previous fingolimod trial to be eligible to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4125 (Actual)
Dates: Start 2010-09-13 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (365):
- United States (33):
  - Novartis Investigative Site, Cullman, Alabama
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Sunrise, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Vero Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Tualatin, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Bristol, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Seattle, Washington
- Argentina (8):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Villa Nueva, Mendoza Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Salta
- Australia (10):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Chatswood, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, North Gosford, New South Wales
  - Novartis Investigative Site, Woodville, South Australia
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Austria (5):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Sankt Pölten
  - Novartis Investigative Site, Vienna
- Belgium (11):
  - Novartis Investigative Site, Fraiture En Condroz, Belgium
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Melsbroek
  - Novartis Investigative Site, Overpelt
  - Novartis Investigative Site, Sijsele
  - Novartis Investigative Site, Sint-Truiden
  - Novartis Investigative Site, Wilrijk
- Brazil (5):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Rio de Janiero, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
- Canada (15):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Nepean, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan
- Czechia (8):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Olomouc, CZE
  - Novartis Investigative Site, Ostrava-Poruba
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Plzen - Lochotin
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Rychnov nad Kněžnou
  - Novartis Investigative Site, Teplice
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
- Egypt (2):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- Novartis Investigative Site, Tallinn, Estonia
- Finland (4):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Seinäjoki
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (16):
  - Novartis Investigative Site, Nancy, Cedex
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poissy
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (91):
  - Novartis Investigative Site, Ostfildern, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Aalen
  - Novartis Investigative Site, Abensberg
  - Novartis Investigative Site, Achim
  - Novartis Investigative Site, Alzenau in Unterfranken
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Honnef
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Bad Neustadt an der Saale
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bogen
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Buchholz
  - Novartis Investigative Site, Buchholz in der Nordheide
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dillingen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Emden
  - Novartis Investigative Site, Emmendingen
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Grevenbroich
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Hennigsdorf
  - Novartis Investigative Site, Herborn
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Ibbenbueren
  - Novartis Investigative Site, Itzehoe
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kaltenkirchen
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Landshut
  - Novartis Investigative Site, Lappersdorf
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lohr a. Main
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nagold
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Neuburg an der Donau
  - Novartis Investigative Site, Neuruppin
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Pforzheim
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Prien am Chiemsee
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Rülzheim
  - Novartis Investigative Site, Schwarzenbruck
  - Novartis Investigative Site, Schwendi
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Sinsheim
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Teupitz
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
  - Novartis Investigative Site, Wendlingen
  - Novartis Investigative Site, Wermsdorf
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Würzburg
- Greece (7):
  - Novartis Investigative Site, Alexandroupoli, Evros
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (9):
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Dublin, Ireland
- Israel (4):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Sefad
- Italy (28):
  - Novartis Investigative Site, Asti, AT
  - Novartis Investigative Site, Acquaviva delle Fonti, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Montichiari, BS
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Fidenza, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Ravenna, RA
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Gallarate, VA
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Viterbo, VT
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Irbid, Jordan
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kuala Lumpur
- Netherlands (10):
  - Novartis Investigative Site, Breda, CK
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Blaricum
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Gouda
  - Novartis Investigative Site, Nieuwegein
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Sittard-Geleen
  - Novartis Investigative Site, Tilburg
- Norway (3):
  - Novartis Investigative Site, Lillehammer
  - Novartis Investigative Site, Molde
  - Novartis Investigative Site, Stavanger
- Novartis Investigative Site, Panama City, Panama
- Peru (3):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, La Perla, Provincia Constitucional del Callao
- Poland (7):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Portugal (5):
  - Novartis Investigative Site, Amadora
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Setúbal
- Romania (3):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Târgu Mureş
- Russia (7):
  - Novartis Investigative Site, Samara, Samara Oblast
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (4):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Trnava
- South Africa (3):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Rosebank
- South Korea (2):
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul
- Spain (11):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santa Cruz de Tenerife
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
- Switzerland (7):
  - Novartis Investigative Site, Aarau
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Carouge
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (11):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Haseki / Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Samsun
  - Novartis Investigative Site, Trabzon
  - Novartis Investigative Site, Yenisehir / Izmir
- United Kingdom (20):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Brighton, East Sussex
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Headington, Oxfordshire
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Dundee
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Essex
  - Novartis Investigative Site, Great Yarmouth
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Northampton
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Poole
  - Novartis Investigative Site, Swindon

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Cohen JA, Tenenbaum N, Bhatt A, Zhang Y, Kappos L. Extended treatment with fingolimod for relapsing multiple sclerosis: the 14-year LONGTERMS study results. Ther Adv Neurol Disord. 2019 Sep 25;12:1756286419878324. doi: 10.1177/1756286419878324. eCollection 2019. PMID 31598139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, multi-center, single treatment arm design allowing patients participating in the fingolimod MS clinical development program to enroll in order to collect additional long-term safety, tolerability, efficacy, and health outcomes data.
Pre-assignment Details: This study had two parts: Part 1, collecting long-term safety, tolerability, efficacy and health outcomes data until all Part 1 end of study (EOS) visits and last follow-up visit; Part 2, collecting limited safety and tolerability data, in a subset of patients who participated in Part 1, and other eligible patients from ongoing fingolimod trials.
Period: Overall Study
Arm/Group | Fingolimod 0.5 mg/Day
Started (All enrolled patients) | 4125
Safety Set (At least one dose of fingolimod in any study and a post-baseline safety assessment) | 4083
Fingolimod Full Analysis Set | 4046
Completed | 3481
Not Completed | 644
Not completed — Adverse Event | 170
Not completed — Abnormal laboratory value(s) | 51
Not completed — Abnormal test procedure result(s) | 3
Not completed — Unsatisfactory therapeutic effect | 112
Not completed — Condition no longer requires study drug | 12
Not completed — Withdrawal by Subject | 144
Not completed — Lost to Follow-up | 50
Not completed — administrative problems | 74
Not completed — Death | 16
Not completed — Protocol Violation | 12

BASELINE CHARACTERISTICS:
Population: Participant Flow and Baseline Characteristics were based on the Enrolled set. Efficacy analyses were based on the Fingolimod Full Analysis Set..
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4125
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (9.05)
Age, Customized [Number; unit: Participants]
  < 18 years | 1
  18 - 30 years | 951
  31 - 40 years | 1497
  41 - 55 years | 1605
  > 55 years | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2933
  Male | 1192
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 3927
  Black | 38
  Asian | 35
  Native American | 11
  Other | 114

OUTCOME MEASURES:

1. Primary Outcome: Parts I and II: Number of Participants With Adverse Events, Serious Adverse Event, and Death
Description: Analysis of absolute and relative frequencies for Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC) to demonstrate that Fingolimod 0.5 mg/day is safe in patients with relapsing forms of Multiple Sclerosis (MS) through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive analysis performed.
Time Frame: Baseline (Part I) to Month 6 Follow-up (Part II), up to 8 years
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4083
Participants
  Adverse Event (AEs) | 2125
  Serious Adverse Events (SAEs) | 515
  Deaths | 16

2. Secondary Outcome: Part I: Aggregate Annualized Relapse Rates (ARR) From First Dose of Fingolimod
Description: Annualized relapse rate (ARR) is defined as the number of all relapses (including both confirmed and unconfirmed relapses) experienced during a specific period of time adjusted to a one-year period. ARR is calculated as follows: (total number of all relapses) / (total number of days in the study for all patients for that specific period of time) x 365.25. Month 0 is the first dose of fingolimod study drug among all studies in which patient participated. Only descriptive analysis performed.
Time Frame: Month 0 (Core Baseline) to End of Follow-up Visit (an average of 162 months)
Population: Fingolimod full analysis set. Only participants with an observed value were considered for the analysis.
Measure: Number; unit: Annual number of relapses per patient
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
Annual number of relapses per patient
  Month 0 to Month 6 | 0.325
  Month 0 to Month 12 | 0.273
  Month 0 to Month 24 | 0.237
  Month 0 to Month 36 | 0.217
  Month 0 to Month 48 | 0.208
  Month 0 to Month 60 | 0.197
  Month 0 to Month 72 | 0.190
  Month 0 to Month 84 | 0.182
  Month 0 to Month 96 | 0.177
  Month 0 to Month 108 | 0.172
  Month 0 to Month 120 | 0.170
  Month 0 to Month 132 | 0.170
  Month 0 to Month 144 | 0.169
  Month 0 to Month 156 | 0.169
  Month 0 to end of Study | 0.166
  Month 0 to end of Follow-up | 0.169

3. Secondary Outcome: Part I: Number of Participants With Relapses (Confirmed and Unconfirmed) From First Dose of Fingolimod
Description: A relapse is defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must be present for at least 24 hours and occur in the absence of fever (<37.5°C) or infection.
  In Study Part One, a relapse must be confirmed by an Expanded Disability Status Scale (EDSS) certified Physician within 7 days of the onset of symptoms. A relapse is confirmed when it is accompanied by an increase of at least half a step (0.5) on the EDSS or an increase of 1 point on two different Functional Systems (FS) of the EDSS or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS). Month 0 is the first dose of fingolimod study drug among all studies in which patient participated. Only descriptive analysis performed.
Time Frame: Month 0 (Core Baseline) to End of Follow-up Visit (an average of 162 months)
Population: Fingolimod full analysis set. Only participants with an observed value were considered for the analysis.
Measure: Number; unit: Participants
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
Participants
  Month 0 to Month 6 | 655
  Month 0 to Month 12 | 992
  Month 0 to Month 24 | 1461
  Month 0 to Month 36 | 1794
  Month 0 to Month 48 | 2127
  Month 0 to Month 60 | 2383
  Month 0 to Month 72 | 2616
  Month 0 to Month 84 | 2793
  Month 0 to Month 96 | 2944
  Month 0 to Month 108 | 3036
  Month 0 to Month 120 | 3063
  Month 0 to Month 132 | 3072
  Month 0 to Month 144 | 3075
  Month 0 to Month 156 | 3079
  Month 0 to end of Study | 2970
  Month 0 to end of Follow-up | 3079

4. Secondary Outcome: Part I: Annualized Rates of New or Newly Enlarging T2 Lesions (ARneT2) Compared With First Dose of Fingolimod
Description: Annualized rate of new/newly enlarging T2 lesions (ARneT2) is defined as the number of new or newly enlarging T2 lesions experienced during a specific period of time adjusted to a one-year period. ARneT2 was calculated as follows: (total number of new/newly enlarging T2 lesions) / (total number of days in the study for all patients for that specific period of time) x 365.25.Month 0 is the first dose of fingolimod study drug among all studies in which patient participated. Only descriptive analysis performed.
Time Frame: Month 0 (Core Baseline) to End of Study (an average of Month 156)
Population: Fingolimod full analysis set. Only participants with an observed value were considered for the analysis.
Measure: Number; unit: Annual number of T2 lesions per patient
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
Annual number of T2 lesions per patient
  Month 0 to Month 3: number analyzed (Participants) | 126
  Month 0 to Month 3 | 12.324
  Month 0 to Month 6: number analyzed (Participants) | 785
  Month 0 to Month 6 | 2.073
  Month 0 to Month 12: number analyzed (Participants) | 1771
  Month 0 to Month 12 | 1.360
  Month 0 to Month 24: number analyzed (Participants) | 1730
  Month 0 to Month 24 | 1.042
  Month 0 to Month 36: number analyzed (Participants) | 1514
  Month 0 to Month 36 | 1.011
  Month 0 to Month 48: number analyzed (Participants) | 1453
  Month 0 to Month 48 | 1.008
  Month 0 to Month 60: number analyzed (Participants) | 1231
  Month 0 to Month 60 | 0.957
  Month 0 to Month 72: number analyzed (Participants) | 1270
  Month 0 to Month 72 | 0.963
  Month 0 to Month 84: number analyzed (Participants) | 1107
  Month 0 to Month 84 | 0.906
  Month 0 to Month 96: number analyzed (Participants) | 578
  Month 0 to Month 96 | 0.813
  Month 0 to Month 108: number analyzed (Participants) | 651
  Month 0 to Month 108 | 0.713
  Month 0 to Month 120: number analyzed (Participants) | 265
  Month 0 to Month 120 | 0.702
  Month 0 to Month 132: number analyzed (Participants) | 52
  Month 0 to Month 132 | 0.659
  Month 0 to Month 144: number analyzed (Participants) | 47
  Month 0 to Month 144 | 0.681
  Month 0 to Month 156: number analyzed (Participants) | 35
  Month 0 to Month 156 | 0.637
  Month 0 to end of study: number analyzed (Participants) | 1320
  Month 0 to end of study | 0.751

5. Secondary Outcome: Part I: Change From First Dose of Fingolimod in Total T2 Lesions Volume
Description: Total volume of T2 lesions was summarized by presenting descriptive statistics for change from first dose of fingolimod baseline values by visit.
Time Frame: Month 3 to End of Study (Study Completion Visit)
Population: Fingolimod full analysis set. Only participants with an observed value were considered for the analysis.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
mm^3
  T2 volume change at Month 3: number analyzed (Participants) | 37
  T2 volume change at Month 3 | -749.5 (5269.04)
  T2 volume change at Month 6: number analyzed (Participants) | 111
  T2 volume change at Month 6 | -207.0 (1385.64)
  T2 volume change at Month 12: number analyzed (Participants) | 1747
  T2 volume change at Month 12 | -55.0 (1700.16)
  T2 volume change at Month 24: number analyzed (Participants) | 1591
  T2 volume change at Month 24 | 16.2 (2009.87)
  T2 volume change at Month 36: number analyzed (Participants) | 1463
  T2 volume change at Month 36 | 235.8 (2519.39)
  T2 volume change at Month 48: number analyzed (Participants) | 1136
  T2 volume change at Month 48 | 875.1 (4145.99)
  T2 volume change at Month 60: number analyzed (Participants) | 1181
  T2 volume change at Month 60 | 1546.3 (4556.51)
  T2 volume change at Month 72: number analyzed (Participants) | 1273
  T2 volume change at Month 72 | 1719.2 (5184.27)
  T2 volume change at Month 84: number analyzed (Participants) | 1053
  T2 volume change at Month 84 | 1635.8 (5075.13)
  T2 volume change at Month 96: number analyzed (Participants) | 569
  T2 volume change at Month 96 | 1303.9 (4712.78)
  T2 volume change at Month 108: number analyzed (Participants) | 648
  T2 volume change at Month 108 | 1562.0 (4654.67)
  T2 volume change at Month 120: number analyzed (Participants) | 261
  T2 volume change at Month 120 | 1393.1 (4908.76)
  T2 volume change at Month 132: number analyzed (Participants) | 50
  T2 volume change at Month 132 | 905.9 (3960.94)
  T2 volume change at Month 144: number analyzed (Participants) | 44
  T2 volume change at Month 144 | 702.7 (3765.80)
  T2 volume change at Month 156: number analyzed (Participants) | 35
  T2 volume change at Month 156 | 274.0 (5784.85)
  T2 volume change at End of Study: number analyzed (Participants) | 1314
  T2 volume change at End of Study | 1588.5 (5157.00)

6. Secondary Outcome: Part I: Change From First Dose of Fingolimod in Total T1 Hypointense Lesions Volume
Description: T1 hypointense lesion (black hole) volume was summarized by presenting descriptive statistics for change from first dose of fingolimod baseline values by visit.
Time Frame: Month 3 to End of Study (Study Completion Visit)
Population: Fingolimod full analysis set. Only participants with an observed value were considered for the analysis.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
mm^3
  T1 volume change at Month 3: number analyzed (Participants) | 12
  T1 volume change at Month 3 | -519.8 (1339.62)
  T1 volume change at Month 12: number analyzed (Participants) | 988
  T1 volume change at Month 12 | 49.1 (718.77)
  T1 volume change at Month 24: number analyzed (Participants) | 1490
  T1 volume change at Month 24 | 64.1 (786.02)
  T1 volume change at Month 36: number analyzed (Participants) | 1348
  T1 volume change at Month 36 | 151.08 (1001.28)
  T1 volume change at Month 48: number analyzed (Participants) | 1023
  T1 volume change at Month 48 | 524.8 (1706.26)
  T1 volume change at Month 60: number analyzed (Participants) | 1068
  T1 volume change at Month 60 | 853.6 (1957.74)
  T1 volume change at Month 72: number analyzed (Participants) | 1175
  T1 volume change at Month 72 | 975.7 (2637.67)
  T1 volume change at Month 84: number analyzed (Participants) | 1012
  T1 volume change at Month 84 | 930.1 (2471.70)
  T1 volume change at Month 96: number analyzed (Participants) | 533
  T1 volume change at Month 96 | 753.4 (1845.63)
  T1 volume change at Month 108: number analyzed (Participants) | 554
  T1 volume change at Month 108 | 628.7 (1922.45)
  T1 volume change at Month 120: number analyzed (Participants) | 172
  T1 volume change at Month 120 | 817.3 (2198.58)
  T1 volume change at Month 132: number analyzed (Participants) | 1
  T1 volume change at Month 132 | 726.7 (NA) — NA: Not estimable due to insufficient number of participants with events
  T1 volume change at End of Study: number analyzed (Participants) | 1236
  T1 volume change at End of Study | 800.6 (2247.27)

7. Secondary Outcome: Part I: Percent Brain Volume Change (PBVC) Relative to First Dose of Fingolimod
Description: Descriptive statistics on percent brain volume change from first dose of fingolimod baseline were presented by visit. A negative change from baseline indicates improvement.
Time Frame: Month 3 to Month 156
Population: Fingolimod full analysis set. Only participants with an observed value were considered for the analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
Percent change
  Percent volume change at Month 3: number analyzed (Participants) | 19
  Percent volume change at Month 3 | -0.19 (0.660)
  Percent volume change at Month 6: number analyzed (Participants) | 758
  Percent volume change at Month 6 | -0.20 (0.801)
  Percent volume change at Month 12: number analyzed (Participants) | 1720
  Percent volume change at Month 12 | -0.36 (0.901)
  Percent volume change at Month 24: number analyzed (Participants) | 1699
  Percent volume change at Month 24 | -0.74 (1.209)
  Percent volume change at Month 36: number analyzed (Participants) | 1480
  Percent volume change at Month 36 | -1.03 (1.541)
  Percent volume change at Month 48: number analyzed (Participants) | 1414
  Percent volume change at Month 48 | -1.44 (1.851)
  Percent volume change at Month 60: number analyzed (Participants) | 1113
  Percent volume change at Month 60 | -1.65 (2.196)
  Percent volume change at Month 72: number analyzed (Participants) | 1151
  Percent volume change at Month 72 | -2.02 (2.514)
  Percent volume change at Month 84: number analyzed (Participants) | 950
  Percent volume change at Month 84 | -2.38 (2.638)
  Percent volume change at Month 96: number analyzed (Participants) | 511
  Percent volume change at Month 96 | -2.41 (2.607)
  Percent volume change at Month 108: number analyzed (Participants) | 593
  Percent volume change at Month 108 | -2.91 (2.863)
  Percent volume change at Month 120: number analyzed (Participants) | 238
  Percent volume change at Month 120 | -3.42 (2.911)
  Percent volume change at Month 132: number analyzed (Participants) | 48
  Percent volume change at Month 132 | -4.61 (2.511)
  Percent volume change at Month 144: number analyzed (Participants) | 45
  Percent volume change at Month 144 | -4.21 (2.778)
  Percent volume change at Month 156: number analyzed (Participants) | 35
  Percent volume change at Month 156 | -4.33 (3.146)

8. Secondary Outcome: Part I: Annualized Rate of Brain Atrophy (ARBA) Relative to First Dose of Fingolimod
Description: The annualized rate of brain volume change is an "averaged annual percentage change" in brain volume. ARBA was calculated as: ARBA = [(SIENA/100+1) ^ (365.25/#days)-1]*100 where SIENA=(Vk/V0-1)*100 and Vk is the brain volume at time k, V0 is the brain volume at time 0 and k is the total number of days in the study for all patients for that specific period of time) × 365.25. Only descriptive analysis performed.
Time Frame: Month 3 to Month 156
Population: Fingolimod full analysis set. Only participants with an observed value were considered for the analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
Ratio
  Month 3: number analyzed (Participants) | 19
  Month 3 | -0.73 (2.834)
  Month 6: number analyzed (Participants) | 758
  Month 6 | -0.39 (1.590)
  Month 12: number analyzed (Participants) | 1720
  Month 12 | -0.35 (0.891)
  Month 24: number analyzed (Participants) | 1699
  Month 24 | -0.37 (0.615)
  Month 36: number analyzed (Participants) | 1480
  Month 36 | -0.35 (0.522)
  Month 48: number analyzed (Participants) | 1414
  Month 48 | -0.37 (0.480)
  Month 60: number analyzed (Participants) | 1113
  Month 60 | -0.34 (0.451)
  Month 72: number analyzed (Participants) | 1151
  Month 72 | -0.35 (0.433)
  Month 84: number analyzed (Participants) | 950
  Month 84 | -0.35 (0.395)
  Month 96: number analyzed (Participants) | 511
  Month 96 | -0.31 (0.340)
  Month 108: number analyzed (Participants) | 593
  Month 108 | -0.33 (0.326)
  Month 120: number analyzed (Participants) | 238
  Month 120 | -0.36 (0.308)
  Month 132: number analyzed (Participants) | 48
  Month 132 | -0.43 (0.240)
  Month 144: number analyzed (Participants) | 45
  Month 144 | -0.36 (0.244)
  Month 156: number analyzed (Participants) | 35
  Month 156 | -0.35 (0.256)

9. Secondary Outcome: Part I: Number of Participants With Confirmed 6-month Disability Progression After First Dose of Fingolimod
Description: Disability progression was defined based on an increase in the EDSS score by 1.5 point for patients with a first dose of fingolimod (FDF) baseline EDSS score of 0, 1 point for patients with FDF baseline EDSS of >=1 and <=5.5, and by 0.5 points for patients with an FDF baseline EDSS>5.5, confirmed after 6 months and all intermediate EDSS assessments. A 6-month confirmed disability progression was defined as a 6-month sustained increase from the reference (potential onset of progression) value in the EDSS scores. i.e., every EDSS score (scheduled or unscheduled) within a 6-month duration after the first progression should meet the progression criteria as specified above. The confirmation could only happen at a scheduled visit and in the absence of a relapse. Only descriptive analysis performed.
Time Frame: Month 12 to Month 156
Population: Fingolimod full analysis set
Measure: Number; unit: Participants
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
Participants
  Month 12 | 212
  Month 24 | 336
  Month 36 | 434
  Month 48 | 519
  Month 60 | 590
  Month 72 | 659
  Month 84 | 714
  Month 96 | 753
  Month 108 | 767
  Month 120 | 772
  Month 132 | 775
  Month 144 | 776
  Month 156 | 777

10. Secondary Outcome: Part I: Number of Participants With Categorized Change From First Dose of Fingolimod in Expanded Disability Status Scale (EDSS) Overall Score
Description: The EDSS is a scale for assessing neurological impairment in MS (Kurtzke 1983) including (1) a series of scores in each of eight functional systems, and (2) the EDSS steps (ranging from 0 (normal) to 10 (death due to MS). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the participant's overall score is categorized as Improvement, Stable or Deterioration.
  If baseline EDSS score is <=5, improvement is indicated by an EDSS score change of <= -1, stable is indicated by an EDSS score change of > -1 and <= 0.5, deterioration is indicated by an EDSS score change of > 0.5; if baseline EDSS score is > 5, improvement is indicated by an EDSS score change of <= -0.5, stable is indicated by an EDSS score change of > -0.5 and <= 0, deterioration is indicated by an EDSS score change of > 0. Only descriptive analysis performed.
Time Frame: Month 3 to Month 6 Follow-up
Population: Fingolimod full analysis set. Only participants with an observed value were considered for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
Participants
  Month 3: number analyzed (Participants) | 3769
  Month 3: Improvement | 374
  Month 3: Stable | 3126
  Month 3: Deterioration | 269
  Month 6: number analyzed (Participants) | 3748
  Month 6: Improvement | 508
  Month 6: Stable | 2900
  Month 6: Deterioration | 340
  Month 9: number analyzed (Participants) | 3211
  Month 9: Improvement | 482
  Month 9: Stable | 2425
  Month 9: Deterioration | 304
  Month 12: number analyzed (Participants) | 2674
  Month 12: Improvement | 422
  Month 12: Stable | 1930
  Month 12: Deterioration | 322
  Month 15: number analyzed (Participants) | 2454
  Month 15: Improvement | 405
  Month 15: Stable | 1764
  Month 15: Deterioration | 285
  Month 18: number analyzed (Participants) | 1977
  Month 18: Improvement | 345
  Month 18: Stable | 1361
  Month 18: Deterioration | 271
  Month 21: number analyzed (Participants) | 2187
  Month 21: Improvement | 376
  Month 21: Stable | 1524
  Month 21: Deterioration | 287
  Month 24: number analyzed (Participants) | 1913
  Month 24: Improvement | 320
  Month 24: Stable | 1299
  Month 24: Deterioration | 294
  Month 27: number analyzed (Participants) | 1854
  Month 27: Improvement | 313
  Month 27: Stable | 1271
  Month 27: Deterioration | 270
  Month 30: number analyzed (Participants) | 1796
  Month 30: Improvement | 305
  Month 30: Stable | 1204
  Month 30: Deterioration | 287
  Month 33: number analyzed (Participants) | 1790
  Month 33: Improvement | 326
  Month 33: Stable | 1172
  Month 33: Deterioration | 292
  Month 36: number analyzed (Participants) | 1662
  Month 36: Improvement | 309
  Month 36: Stable | 1065
  Month 36: Deterioration | 288
  Month 39: number analyzed (Participants) | 1575
  Month 39: Improvement | 284
  Month 39: Stable | 1015
  Month 39: Deterioration | 276
  Month 42: number analyzed (Participants) | 1517
  Month 42: Improvement | 282
  Month 42: Stable | 948
  Month 42: Deterioration | 287
  Month 45: number analyzed (Participants) | 1382
  Month 45: Improvement | 244
  Month 45: Stable | 875
  Month 45: Deterioration | 263
  Month 48: number analyzed (Participants) | 1352
  Month 48: Improvement | 250
  Month 48: Stable | 838
  Month 48: Deterioration | 264
  Month 51: number analyzed (Participants) | 1275
  Month 51: Improvement | 244
  Month 51: Stable | 784
  Month 51: Deterioration | 247
  Month 54: number analyzed (Participants) | 1295
  Month 54: Improvement | 256
  Month 54: Stable | 788
  Month 54: Deterioration | 251
  Month 57: number analyzed (Participants) | 1140
  Month 57: Improvement | 201
  Month 57: Stable | 694
  Month 57: Deterioration | 245
  Month 60: number analyzed (Participants) | 986
  Month 60: Improvement | 175
  Month 60: Stable | 577
  Month 60: Deterioration | 234
  Month 63: number analyzed (Participants) | 913
  Month 63: Improvement | 182
  Month 63: Stable | 540
  Month 63: Deterioration | 191
  Month 66: number analyzed (Participants) | 880
  Month 66: Improvement | 165
  Month 66: Stable | 499
  Month 66: Deterioration | 216
  Month 69: number analyzed (Participants) | 852
  Month 69: Improvement | 156
  Month 69: Stable | 503
  Month 69: Deterioration | 193
  Month 72: number analyzed (Participants) | 789
  Month 72: Improvement | 143
  Month 72: Stable | 440
  Month 72: Deterioration | 206
  Month 75: number analyzed (Participants) | 794
  Month 75: Improvement | 156
  Month 75: Stable | 437
  Month 75: Deterioration | 201
  Month 78: number analyzed (Participants) | 760
  Month 78: Improvement | 136
  Month 78: Stable | 398
  Month 78: Deterioration | 226
  Month 81: number analyzed (Participants) | 823
  Month 81: Improvement | 150
  Month 81: Stable | 456
  Month 81: Deterioration | 217
  Month 84: number analyzed (Participants) | 746
  Month 84: Improvement | 132
  Month 84: Stable | 407
  Month 84: Deterioration | 207
  Month 87: number analyzed (Participants) | 824
  Month 87: Improvement | 147
  Month 87: Stable | 450
  Month 87: Deterioration | 227
  Month 90: number analyzed (Participants) | 737
  Month 90: Improvement | 120
  Month 90: Stable | 413
  Month 90: Deterioration | 204
  Month 93: number analyzed (Participants) | 716
  Month 93: Improvement | 143
  Month 93: Stable | 386
  Month 93: Deterioration | 187
  Month 96: number analyzed (Participants) | 678
  Month 96: Improvement | 117
  Month 96: Stable | 375
  Month 96: Deterioration | 186
  Month 99: number analyzed (Participants) | 594
  Month 99: Improvement | 110
  Month 99: Stable | 325
  Month 99: Deterioration | 159
  Month 102: number analyzed (Participants) | 531
  Month 102: Improvement | 94
  Month 102: Stable | 283
  Month 102: Deterioration | 154
  Month 105: number analyzed (Participants) | 495
  Month 105: Improvement | 103
  Month 105: Stable | 261
  Month 105: Deterioration | 131
  Month 108: number analyzed (Participants) | 512
  Month 108: Improvement | 87
  Month 108: Stable | 287
  Month 108: Deterioration | 138
  Month 111: number analyzed (Participants) | 373
  Month 111: Improvement | 74
  Month 111: Stable | 198
  Month 111: Deterioration | 101
  Month 114: number analyzed (Participants) | 305
  Month 114: Improvement | 45
  Month 114: Stable | 181
  Month 114: Deterioration | 79
  Month 117: number analyzed (Participants) | 177
  Month 117: Improvement | 31
  Month 117: Stable | 94
  Month 117: Deterioration | 52
  Month 120: number analyzed (Participants) | 149
  Month 120: Improvement | 19
  Month 120: Stable | 88
  Month 120: Deterioration | 42
  Month 123: number analyzed (Participants) | 66
  Month 123: Improvement | 9
  Month 123: Stable | 36
  Month 123: Deterioration | 21
  Month 126: number analyzed (Participants) | 85
  Month 126: Improvement | 14
  Month 126: Stable | 45
  Month 126: Deterioration | 26
  Month 129: number analyzed (Participants) | 36
  Month 129: Improvement | 6
  Month 129: Stable | 18
  Month 129: Deterioration | 12
  Month 132: number analyzed (Participants) | 68
  Month 132: Improvement | 11
  Month 132: Stable | 36
  Month 132: Deterioration | 21
  Month 135: number analyzed (Participants) | 36
  Month 135: Improvement | 5
  Month 135: Stable | 19
  Month 135: Deterioration | 12
  Month 138: number analyzed (Participants) | 67
  Month 138: Improvement | 10
  Month 138: Stable | 39
  Month 138: Deterioration | 18
  Month 141: number analyzed (Participants) | 36
  Month 141: Improvement | 6
  Month 141: Stable | 18
  Month 141: Deterioration | 12
  Month 144: number analyzed (Participants) | 56
  Month 144: Improvement | 7
  Month 144: Stable | 30
  Month 144: Deterioration | 19
  Month 147: number analyzed (Participants) | 42
  Month 147: Improvement | 6
  Month 147: Stable | 21
  Month 147: Deterioration | 15
  Month 150: number analyzed (Participants) | 44
  Month 150: Improvement | 7
  Month 150: Stable | 22
  Month 150: Deterioration | 15
  Month 153: number analyzed (Participants) | 32
  Month 153: Improvement | 8
  Month 153: Stable | 16
  Month 153: Deterioration | 8
  Month 156: number analyzed (Participants) | 17
  Month 156: Improvement | 3
  Month 156: Stable | 9
  Month 156: Deterioration | 5
  Month 159: number analyzed (Participants) | 9
  Month 159: Improvement | 1
  Month 159: Stable | 2
  Month 159: Deterioration | 6
  Month 162: number analyzed (Participants) | 2
  Month 162: Improvement | 0
  Month 162: Stable | 1
  Month 162: Deterioration | 1
  End of study: number analyzed (Participants) | 3814
  End of study: Improvement | 610
  End of study: Stable | 2419
  End of study: Deterioration | 785
  Month 3 follow-up: number analyzed (Participants) | 1491
  Month 3 follow-up: Improvement | 203
  Month 3 follow-up: Stable | 907
  Month 3 follow-up: Deterioration | 381
  Month 6 follow-up: number analyzed (Participants) | 228
  Month 6 follow-up: Improvement | 29
  Month 6 follow-up: Stable | 111
  Month 6 follow-up: Deterioration | 88

11. Secondary Outcome: Part I: Change From First Dose of Fingolimod in Expanded Disability Status Scale (EDSS)
Description: The EDSS is a scale for assessing neurological impairment in MS (Kurtzke 1983) including (1) a series of scores in each of eight functional systems, and (2) the EDSS steps (ranging from 0 (normal) to 10 (death due to MS). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the participant's overall score is determined between 0 to 10. A negative change from baseline indicates improvement. Only descriptive analysis performed.
Time Frame: Month 0 (Core Baseline) to End of Follow-up Visit (an average of 162 months)
Population: Fingolimod full analysis set. Only participants with an observed value were considered for the analysis.
Measure: Mean (Standard Deviation); unit: EDDS Overall Score
Arm/Group | Fingolimod 0.5 mg/Day
Number analyzed (Participants) | 4046
EDDS Overall Score
  Baseline (BL): number analyzed (Participants) | 4042
  Baseline (BL) | 2.39 (1.452)
  Change from BL at Month 3: number analyzed (Participants) | 3769
  Change from BL at Month 3 | -0.06 (0.638)
  Change from BL at Month 6: number analyzed (Participants) | 3748
  Change from BL at Month 6 | -0.07 (0.716)
  Change from BL at Month 9: number analyzed (Participants) | 3211
  Change from BL at Month 9 | -0.09 (0.750)
  Change from BL at Month 12: number analyzed (Participants) | 2674
  Change from BL at Month 12 | -0.07 (0.815)
  Change from BL at Month 15: number analyzed (Participants) | 2454
  Change from BL at Month 15 | -0.08 (0.814)
  Change from BL at Month 18: number analyzed (Participants) | 1977
  Change from BL at Month 18 | -0.05 (0.890)
  Change from BL at Month 21: number analyzed (Participants) | 2187
  Change from BL at Month 21 | -0.08 (0.876)
  Change from BL at Month 24: number analyzed (Participants) | 1913
  Change from BL at Month 24 | -0.01 (0.916)
  Change from BL at Month 27: number analyzed (Participants) | 1854
  Change from BL at Month 27 | -0.03 (0.932)
  Change from BL at Month 30: number analyzed (Participants) | 1796
  Change from BL at Month 30 | -0.00 (0.935)
  Change from BL at Month 33: number analyzed (Participants) | 1790
  Change from BL at Month 33 | -0.02 (0.951)
  Change from BL at Month 36: number analyzed (Participants) | 1662
  Change from BL at Month 36 | 0.01 (0.997)
  Change from BL at Month 39: number analyzed (Participants) | 1575
  Change from BL at Month 39 | 0.02 (0.963)
  Change from BL at Month 42: number analyzed (Participants) | 1517
  Change from BL at Month 42 | 0.04 (1.015)
  Change from BL at Month 45: number analyzed (Participants) | 1382
  Change from BL at Month 45 | 0.06 (1.006)
  Change from BL at Month 48: number analyzed (Participants) | 1352
  Change from BL at Month 48 | 0.06 (1.063)
  Change from BL at Month 51: number analyzed (Participants) | 1275
  Change from BL at Month 51 | 0.06 (1.071)
  Change from BL at Month 54: number analyzed (Participants) | 1295
  Change from BL at Month 54 | 0.04 (1.120)
  Change from BL at Month 57: number analyzed (Participants) | 1140
  Change from BL at Month 57 | 0.09 (1.077)
  Change from BL at Month 60: number analyzed (Participants) | 986
  Change from BL at Month 60 | 0.17 (1.144)
  Change from BL at Month 63: number analyzed (Participants) | 913
  Change from BL at Month 63 | 0.08 (1.123)
  Change from BL at Month 66: number analyzed (Participants) | 880
  Change from BL at Month 66 | 0.15 (1.220)
  Change from BL at Month 69: number analyzed (Participants) | 852
  Change from BL at Month 69 | 0.14 (1.116)
  Change from BL at Month 72: number analyzed (Participants) | 789
  Change from BL at Month 72 | 0.22 (1.205)
  Change from BL at Month 75: number analyzed (Participants) | 794
  Change from BL at Month 75 | 0.13 (1.159)
  Change from BL at Month 78: number analyzed (Participants) | 760
  Change from BL at Month 78 | 0.28 (1.259)
  Change from BL at Month 81: number analyzed (Participants) | 823
  Change from BL at Month 81 | 0.18 (1.158)
  Change from BL at Month 84: number analyzed (Participants) | 746
  Change from BL at Month 84 | 0.25 (1.236)
  Change from BL at Month 87: number analyzed (Participants) | 824
  Change from BL at Month 87 | 0.24 (1.206)
  Change from BL at Month 90: number analyzed (Participants) | 737
  Change from BL at Month 90 | 0.29 (1.282)
  Change from BL at Month 93: number analyzed (Participants) | 716
  Change from BL at Month 93 | 0.18 (1.219)
  Change from BL at Month 96: number analyzed (Participants) | 678
  Change from BL at Month 96 | 0.31 (1.355)
  Change from BL at Month 99: number analyzed (Participants) | 594
  Change from BL at Month 99 | 0.18 (1.220)
  Change from BL at Month 102: number analyzed (Participants) | 531
  Change from BL at Month 102 | 0.30 (1.332)
  Change from BL at Month 105: number analyzed (Participants) | 495
  Change from BL at Month 105 | 0.21 (1.320)
  Change from BL at Month 108: number analyzed (Participants) | 512
  Change from BL at Month 108 | 0.28 (1.270)
  Change from BL at Month 111: number analyzed (Participants) | 373
  Change from BL at Month 111 | 0.24 (1.343)
  Change from BL at Month 114: number analyzed (Participants) | 305
  Change from BL at Month 114 | 0.30 (1.258)
  Change from BL at Month 117: number analyzed (Participants) | 177
  Change from BL at Month 117 | 0.35 (1.389)
  Change from BL at Month 120: number analyzed (Participants) | 149
  Change from BL at Month 120 | 0.40 (1.271)
  Change from BL at Month 123: number analyzed (Participants) | 66
  Change from BL at Month 123 | 0.60 (1.302)
  Change from BL at Month 126: number analyzed (Participants) | 85
  Change from BL at Month 126 | 0.38 (1.441)
  Change from BL at Month 129: number analyzed (Participants) | 36
  Change from BL at Month 129 | 0.40 (1.448)
  Change from BL at Month 132: number analyzed (Participants) | 68
  Change from BL at Month 132 | 0.40 (1.450)
  Change from BL at Month 135: number analyzed (Participants) | 36
  Change from BL at Month 135 | 0.51 (1.519)
  Change from BL at Month 138: number analyzed (Participants) | 67
  Change from BL at Month 138 | 0.42 (1.527)
  Change from BL at Month 141: number analyzed (Participants) | 36
  Change from BL at Month 141 | 0.54 (1.509)
  Change from BL at Month 144: number analyzed (Participants) | 56
  Change from BL at Month 144 | 0.60 (1.553)
  Change from BL at Month 147: number analyzed (Participants) | 42
  Change from BL at Month 147 | 0.67 (1.640)
  Change from BL at Month 150: number analyzed (Participants) | 44
  Change from BL at Month 150 | 0.44 (1.483)
  Change from BL at Month 153: number analyzed (Participants) | 32
  Change from BL at Month 153 | 0.23 (1.534)
  Change from BL at Month 156: number analyzed (Participants) | 17
  Change from BL at Month 156 | 0.26 (1.427)
  Change from BL at Month 159: number analyzed (Participants) | 9
  Change from BL at Month 159 | 1.17 (1.369)
  Change from BL at Month 162: number analyzed (Participants) | 2
  Change from BL at Month 162 | 0.75 (1.061)
  Change from BL at End of study: number analyzed (Participants) | 3814
  Change from BL at End of study | 0.14 (1.108)
  Change from BL at Month 3 follow-up: number analyzed (Participants) | 1491
  Change from BL at Month 3 follow-up | 0.29 (1.248)
  Change from BL at Month 6 follow-up: number analyzed (Participants) | 228
  Change from BL at Month 6 follow-up | 0.56 (1.487)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment in Study Part I until end of study treatment in Study Part II plus 6 weeks post treatment, up to a maximum duration of 8 years.
Arm/Group | Fingolimod 0.5 mg/Day
All-Cause Mortality (participants affected / at risk) | 16/4083
Serious Adverse Events (participants affected / at risk) | 515/4083
Other Adverse Events (participants affected / at risk) | 2125/4083
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg/Day (N=4083)
Anaemia (Blood and lymphatic system disorders) | 3
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 6
Atrioventricular block first degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Cardiovascular insufficiency (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Pericarditis (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 3
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 1
Congenital cytomegalovirus infection (Congenital, familial and genetic disorders) | 1
Congenital knee dislocation (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 4
Hyperprolactinaemia (Endocrine disorders) | 1
Thyroid mass (Endocrine disorders) | 1
Photophobia (Eye disorders) | 1
Retinal detachment (Eye disorders) | 2
Retinal haemorrhage (Eye disorders) | 1
Retinal vein thrombosis (Eye disorders) | 1
Abdominal adhesions (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 4
Barrett's oesophagus (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 3
Irritable bowel syndrome (Gastrointestinal disorders) | 2
Large intestine polyp (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Rectal polyp (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Death (General disorders) | 2
Death neonatal (General disorders) | 1
Fat tissue increased (General disorders) | 1
Fatigue (General disorders) | 5
Gait disturbance (General disorders) | 2
Hernia (General disorders) | 1
Hypothermia (General disorders) | 2
Influenza like illness (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 5
Vascular stent stenosis (General disorders) | 1
Biliary colic (Hepatobiliary disorders) | 5
Biliary cyst (Hepatobiliary disorders) | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 4
Cholecystitis chronic (Hepatobiliary disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 10
Drug-induced liver injury (Hepatobiliary disorders) | 2
Hepatitis acute (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1
Immunodeficiency (Immune system disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Abdominal sepsis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 10
Appendicitis perforated (Infections and infestations) | 2
Bartholin's abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 6
Cystitis (Infections and infestations) | 1
Dermatitis infected (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 2
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Hepatitis A (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 2
Hepatitis E (Infections and infestations) | 1
Herpes simplex encephalitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 9
Herpes zoster infection neurological (Infections and infestations) | 1
Histoplasmosis (Infections and infestations) | 1
Infected dermal cyst (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Injection site abscess (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Meningitis cryptococcal (Infections and infestations) | 1
Meningoencephalitis herpetic (Infections and infestations) | 1
Orchitis (Infections and infestations) | 2
Pelvic inflammatory disease (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 14
Pneumonia bacterial (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Renal abscess (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Salpingitis (Infections and infestations) | 1
Salpingo-oophoritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Spermatic cord funiculitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 14
Urinary tract infection enterococcal (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Viraemia (Infections and infestations) | 1
Viral diarrhoea (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Vulval abscess (Infections and infestations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 6
Arthropod bite (Injury, poisoning and procedural complications) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 2
Foot fracture (Injury, poisoning and procedural complications) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
Joint injury (Injury, poisoning and procedural complications) | 1
Kidney contusion (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 2
Meniscus injury (Injury, poisoning and procedural complications) | 2
Multiple injuries (Injury, poisoning and procedural complications) | 1
Muscle injury (Injury, poisoning and procedural complications) | 1
Near drowning (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 5
Skull fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 4
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Traumatic spinal cord compression (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 3
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Vaginal laceration (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2
Hepatic enzyme increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Weight decreased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Amyotrophy (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Lateral patellar compression syndrome (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 30
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone giant cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
Altered state of consciousness (Nervous system disorders) | 2
Brain hypoxia (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Cauda equina syndrome (Nervous system disorders) | 1
Central nervous system lesion (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebral venous thrombosis (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Demyelination (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 8
Facial spasm (Nervous system disorders) | 1
Fine motor skill dysfunction (Nervous system disorders) | 1
Focal dyscognitive seizures (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hemianopia homonymous (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hyperaesthesia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 3
Lacunar infarction (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 2
Multiple sclerosis (Nervous system disorders) | 3
Multiple sclerosis relapse (Nervous system disorders) | 34
Muscle spasticity (Nervous system disorders) | 1
Myelitis transverse (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 2
Optic neuritis (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 2
Partial seizures (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 1
Secondary progressive multiple sclerosis (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 3
Spinal cord compression (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 4
Tension headache (Nervous system disorders) | 1
Thrombotic stroke (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 3
Trigeminal neuralgia (Nervous system disorders) | 3
Uhthoff's phenomenon (Nervous system disorders) | 1
Ulnar nerve palsy (Nervous system disorders) | 1
Wernicke's encephalopathy (Nervous system disorders) | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 10
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1
Device dislocation (Product Issues) | 1
Acute stress disorder (Psychiatric disorders) | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 2
Aggression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Bipolar I disorder (Psychiatric disorders) | 2
Completed suicide (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 9
Drug dependence (Psychiatric disorders) | 1
Eating disorder (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 2
Mania (Psychiatric disorders) | 3
Mental disorder (Psychiatric disorders) | 2
Panic attack (Psychiatric disorders) | 2
Persecutory delusion (Psychiatric disorders) | 1
Personality change (Psychiatric disorders) | 1
Personality change due to a general medical condition (Psychiatric disorders) | 1
Psychogenic seizure (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Somatic symptom disorder (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 5
Suicide attempt (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Calculus urinary (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 3
Renal haemorrhage (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Adnexa uteri cyst (Reproductive system and breast disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Breast calcifications (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 7
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 3
Ovarian cyst (Reproductive system and breast disorders) | 4
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1
Uterine cyst (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 3
Uterine polyp (Reproductive system and breast disorders) | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Erythema annulare (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Abortion induced (Surgical and medical procedures) | 1
Aneurysm (Vascular disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 4
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Hypoperfusion (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Peripheral venous disease (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1
Venous stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg/Day (N=4083)
Lymphopenia (Blood and lymphatic system disorders) | 219
Fatigue (General disorders) | 232
Bronchitis (Infections and infestations) | 214
Influenza (Infections and infestations) | 275
Nasopharyngitis (Infections and infestations) | 706
Upper respiratory tract infection (Infections and infestations) | 346
Urinary tract infection (Infections and infestations) | 335
Hypercholesterolaemia (Metabolism and nutrition disorders) | 212
Arthralgia (Musculoskeletal and connective tissue disorders) | 208
Back pain (Musculoskeletal and connective tissue disorders) | 279
Headache (Nervous system disorders) | 348
Depression (Psychiatric disorders) | 205
Hypertension (Vascular disorders) | 243

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT01201356/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT01201356/SAP_001.pdf